CLINICAL TRIAL: NCT05647083
Title: The Effect of Massage on Diabetic Foot Risk, HbA1c and Physiological Parameters in People With Type 2 Diabetes
Brief Title: The Effect of Massage on Diabetic Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Elif Gencer Sendur, Associate Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BAIBU-SBF-EGS-2
Record Dates: First submitted 2022-11-21; First posted 2022-12-12 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2; Peripheral Neuropathy
Keywords: massage; glycemic control; diabetic foot risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Peripheral Nervous System Diseases | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A total of 24 massage sessions will be applied to the intervention group, 2 times a week during the 12-week working period. Sesame oil will be used as the main oil in the massage application. Massage times are recommended as 10-15 minutes for upper extremity massage and 15-20 minutes for lower extremity massage.
  Interventions: Other: Massage therapy
- Control group (No Intervention): Participants in the control group will continue their medical treatment protocols and massage will not be applied. Measurement tools and physiological measurements will be evaluated at the frequency specified in the intervention group, using the same measurement tools and the same measurement methods.

INTERVENTIONS:
Other: Massage therapy — Classical massage will be applied to the hands and feet, which is expected to take an average of 30 minutes.
  Arms: Intervention group

SUMMARY:
This research aims to investigate the effect of massage on diabetic foot risk, HbA1c and physiological parameters in individuals with type 2 diabetes. This randomized controlled experimental design will be carried out in Bolu Izzet Baysal State Hospital Köroğlu Unit Internal Medicine Polyclinic and Internal Medicine Service. According to power analysis, the minimum sample size was determined as 60 people, 30 of which were in the intervention group and 30 in the control group. Data collection tools include "Peripheral Neuropathy Sign and Symptom Score", "Ankle-Brachial Index (ABI)", "Glycemic Control Assessment (HbA1c)", "Physiological Parameters (blood pressure, heart rate and oxygen saturation)", "Inlow's 60-second Diabetic Food Screen". A total of 24 massage sessions will be applied to the intervention group, 2 times a week during the 12-week working period. Participants in the control group will continue their medical treatment protocols and massage will not be applied.

ELIGIBILITY:
Inclusion Criteria:

* Being between 30-75 years old,
* Diagnosed with diabetes at least 6 months ago,
* Absence of irritation, ulceration in the areas where the massage will be applied (hands, feet and legs),
* No problem in verbal communication,
* Being able to speak Turkish,
* No diagnosis of psychiatric disease,
* Absence of amputation in the upper and lower extremities,
* Having HbA1c test results in the last 1 week,
* Not having had Covid-19 in the last 6 months
* No experience of massage application in the last 1 month
* Willingness to participate in the research

Exclusion Criteria:

* Presence of diabetic ulcer and foot wound,
* Irritation and ulceration in the areas where the massage will be applied (hands, feet and legs),
* Having problems in verbal communication,
* Not being able to speak Turkish,
* Having a diagnosis of psychiatric illness.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Means of Peripheral Neuropathy Sign and Symptom Score | Change from baseline Neuropathy score at 3 months
  Peripheral neuropathy consists of two parts: symptom and symptom score. For the peripheral neuropathy symptom score;
  * Discomfort they feel in their feet,
  * Location of complaints,
  * The presence of complaints increases at night,
  * Time of occurrence of complaints and
  * 5 questions will be asked about how the complaints decreased. Peripheral neuropathy symptom score obtained from 5 questions was 0-2 points, "normal"; 3-4 points, "mild neuropathy"; 5-6 points, "moderate neuropathy"; A score of 7-9 will be considered "severe neuropathy".
  For peripheral neuropathy finding score; It will be determined based on four parameters including 1. Vibration sense, 2. Pimpiric test, 3. Achille tendon reflex, 4. Protective sensory examination
Means of Ankle-Brachial Index Score | Change from baseline Ankle-Brachial Index score at 3 months
  It is calculated by dividing the tibialis posterior pressure by the brachial arterial pressure. The highest of the four measurements at the ankles and feet is divided by the two higher brachial measurements. The normal value is close to 1.
Means of HbA1c (%) | Change from baseline HbA1c score at 3 months
  HbA1c values of the participants will be monitored as a glycemic control parameter. The HbA1c value will be evaluated at baseline and 3 months later, as it represents the three-month average blood glucose value. For the measurement of HbA1c, the test results within the last week will be taken from the participants at the beginning and a blood sample will be taken into ethylenediaminetetraacetic acid (EDTA) coated tubes (2 mL whole) by a nurse three months later.
Means of systolic blood pressure (mmHg) | Change from baseline systolic blood pressure at 3 months
  It will be measured by the researcher with a manual measurement tool.
Means of diastolic blood pressure (mmHg) | Change from baseline diastolic blood pressure at 3 months
  It will be measured by the researcher with a manual measurement tool.
Means of heart rate (/minutes) | Change from baseline heart rate at 3 months
  It will be measured by the researcher with a pulse oximeter.
Means of oxygen saturation (%) | Change from baseline oxygen saturation at 3 months
  It will be measured by the researcher with a pulse oximeter.
Means of diabetic foot risk score | Change from baseline diabetic foot risk score at 3 months
  "Inlow's 60-second Diabetic Food Screen" form will be used in diabetes foot risk assessment. Diabetic foot examination consists of 12 parameters. Skin Assessment, Evaluation of Nail Structure, deformity, Evaluation of the Shoe, Heat Evaluation - Being Cold, Heat Evaluation - Being Hot, Range of Motion Evaluation, Sensory Evaluation, Sensory Evaluation (Assessment with questions directed to individuals), Evaluation of Pedal Pulses, Dependent Rubor Evaluation, Evaluation of Erythema (Redness). The minimum score to be taken from the foot examination form is evaluated as 0 and the maximum score as 23 points. The higher the score, the higher the risk of diabetic foot.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gençer Şendur, MSC, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Provincial Health Directorate Bolu Izzet Baysal State Hospital, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No